CLINICAL TRIAL: NCT05294367
Title: Pilot Feasibility Trial of Dietary and Topical Magnesium Replacement or Supplementation in Patients With Lymphoma
Brief Title: Dietary and Topical Magnesium Replacement or Supplementation in Patients With Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LS200801; NCI-2022-00602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-005406 (Other: Mayo Clinic Institutional Review Board); P50CA097274 (NIH)
Record Dates: First submitted 2022-03-03; First posted 2022-03-24 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cycle 1 (Experimental): Participants consume magnesium rich foods PO daily for 28 days.
  Interventions: Other: Quality-of-Life Assessment; Behavioral: Special Diet Therapy
- Cycle 2, Arm I (Experimental): Participants continue consuming magnesium rich foods PO daily and apply Ancient Minerals Magnesium Lotion topically daily for 28 days.
  Interventions: Drug: Magnesium Chloride-based Lotion; Other: Quality-of-Life Assessment; Behavioral: Special Diet Therapy
- Cycle 2, Arm II (Experimental): Participants continue consuming magnesium rich foods PO daily for 28 days.
  Interventions: Other: Quality-of-Life Assessment; Behavioral: Special Diet Therapy

INTERVENTIONS:
Drug: Magnesium Chloride-based Lotion — Given topically
  Other Names: Ancient Minerals Magnesium Lotion; Magnesium Chloride Lotion
  Arms: Cycle 2, Arm I
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Behavioral: Special Diet Therapy — Consume magnesium rich foods
  Other Names: DIET

SUMMARY:
This early phase I trial investigates the effect of dietary and topical magnesium replacement on magnesium blood levels in patients with lymphoma. Magnesium is an element in the body that is important to cell health. The body cannot make magnesium and it typically comes from the food we eat. In patients who are ill, magnesium is often replaced intravenously (IV) through a vein or by mouth. This study may help researchers find out if being on a magnesium rich diet and using a magnesium lotion on the skin helps to keep magnesium blood levels in an ideal range. This study also investigates side effects and quality of life when receiving different forms of magnesium.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess if dietary replacement with magnesium rich foods and topical magnesium replacement improves serum magnesium levels in patients with a history of a lymphoproliferative disorder, not on active myelosuppressive chemotherapy, and have a serum magnesium levels 1.5 - 1.9 mg/dL.

SECONDARY OBJECTIVES:

I. Evaluate the compliance of a diet rich in magnesium as well as compliance with topical magnesium replacement in lymphoma patients who have completed therapy and are in remission.

II. Assess feasibility of enrolling patients with a history of lymphoproliferative disorder, not on active treatment with low magnesium levels.

III. Assess tolerability and toxicity of a magnesium rich diet with and without topical magnesium replacement.

EXPLORATORY OBJECTIVES:

I. Assess quality of life in patients receiving magnesium replacement with diet and/or topical magnesium.

II. Evaluate whether magnesium replacement strategies are equally effective between ethnicities.

OUTLINE:

CYCLE 1: Participants consume magnesium rich foods orally (PO) daily for 28 days.

CYCLE 2: Participants with a magnesium level between 1.5-2.1 mg/dL at the end of cycle 1 are assigned to Arm I. Patients with a magnesium level between 2.2-2.3 mg/dL at the end of cycle 1 are assigned to Arm II. Patients with a magnesium level < 1.5 mg/dL at the end of cycle 1 go off study.

ARM I: Participants continue consuming magnesium rich foods PO daily and apply Ancient Minerals Magnesium Lotion topically daily for 28 days.

ARM II: Participants continue consuming magnesium rich foods PO daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION - INCLUSION CRITERIA:

* Age >= 18 years
* Currently have or have had in the past the diagnosis of any type of lymphoma
* If previously treated, the patient must be off myelosuppressive chemotherapy with no planned chemotherapy for >= 2 months. Patients with lymphoproliferative disorders being observed (i.e., never treated) or those on rituximab (or equivalent) maintenance or chronic oral therapies such as BTK inhibitors, venetoclax, tazemetostat, or corticosteroids are also eligible
* Able to eat a full range of solid food and liquids and tolerate seeds/nuts
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1, or 2
* Provide written informed consent
* Able to recollect dietary intake for the prior 24 hours in order to complete a one-day food record with assistance from a dietitian at each study visit
* Willing to be seen at the enrolling institution at baseline, and at 4 weeks and 8 weeks (end of treatment) in person or by video/phone
* Willing to have a blood magnesium checked every 2 weeks x 4 at any Mayo Clinic site
* Ability to complete questionnaire(s) by themselves or with assistance

REGISTRATION - INCLUSION CRITERIA:

* Magnesium level of 1.5 - 1.9 mg/dL (obtained =< 5 days prior to registration)

Exclusion Criteria:

PRE-REGISTRATION - EXCLUSION CRITERIA:

* Cannot eat normal table food by mouth. NOTE: Patients with any form of feeding tube or a swallowing disorder are not eligible
* Have taken dedicated magnesium supplements (i.e. magnesium oxide) or intravenous (IV) magnesium =< 28 days prior to pre-registration. Note: If patient is already on a multivitamin containing -magnesium, they may be enrolled, but the brand should not be changed during the 8 weeks on study
* Co-morbid systemic illnesses such as active infection or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients with significant gut malabsorptive conditions (such as inflammatory bowel disease or others at the discretion of the investigator) will be excluded as well as patients with chronic kidney disease stage 3b or greater (estimated glomerular filtration rate [eGFR] < 45)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent for lymphoma or any other disease
* Active other malignancy requiring treatment that would interfere with the assessments of this study
* Major surgery other than diagnostic surgery =< 4 weeks prior to pre-registration
* Have an allergy to nuts
* Patients with active skin lymphoma or rashes that would preclude lotion testing
* Have taken antibiotics =< 7 days prior to pre-registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in serum magnesium levels | Baseline up to 2 cycles (56 days)
  Will be defined as an increase in magnesium levels of at least 0.2 mg/dL from baseline level or an increase in magnesium level to 2.0 - 2.3 mg/dL at any time after the beginning of replacement.

SECONDARY OUTCOMES:
Feasibility of patient enrollment | Baseline up to 2 cycles (56 days)
  Will be assessed by the percentage of patients that pre-register who continue on to register for the study. Reasons for pre-registering but not continuing on to registration will be summarized descriptively.
Tolerability and Toxicity Assessment | Up to 56 days
  Tolerability and toxicity will be assessed by evaluating the number of days the diet was not properly followed. This will be summarized descriptively.
Incidence of adverse events | Up to 56 days
  Assess the number of doses of topical magnesium replacement missed due to adverse events. Reasons for missed doses will be summarized descriptively.
Patient compliance | Up to 56 days
  Patient compliance with a diet rich in magnesium as well as compliance with topical magnesium replacement will be assessed by evaluating patient medication logs and meal logs. For the magnesium rich diet, a scoring points system will be utilized, where the goal is to achieve 10 points of magnesium in the diet each day. Compliance with the magnesium diet will be defined as meeting at least 7 points daily. For the topical magnesium replacement, the goal is to apply 6 pumps of the lotion daily. Compliance with the topical magnesium replacement will be defined as at least 5 pumps daily. The number of days met for the magnesium rich diet and topical magnesium replacement will be evaluated and summarized descriptively.

OTHER OUTCOMES:
Patient Medication Quality of Life Assessment | At baseline, 28 days, and 56 days
  Will be summarized descriptively and changes across time will be explored by patient completing the Quality of Life Assessment Questionairre.
Relationship between race/ethnicity and differences in diet and serum magnesium levels | Up to 56 days
  Will be assessed to evaluate whether magnesium replacement strategies are equally effective between racial/ethnic groups. The percentage of patients who achieve an improvement in magnesium levels from baseline will be evaluated in each racial/ethnic group to assess whether differences may exist.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials